CLINICAL TRIAL: NCT01562977
Title: Prospective, Open-label, Multicentric, ph. II Study of R-GemOx and Dexametasone in Patients With Agressive Lymphomas Refractory or Relapsed to Previous Treatment and Non Eligible for High-dose Chemotherapy Followed by Autologous Stem Cell Transplanted
Brief Title: Study to Evaluate Efficacy and Tolerance of R-GemOx in DLBCL and MCL
Acronym: RGemOx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Principal Investigator, Ana Mendez Lopez, Sponsor's secretary, Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEL-TAMO/R-GemOx-08-04/v2
Record Dates: First submitted 2011-07-18; First posted 2012-03-26 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Aggressive Lymphoma; Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Rituximab; Gemcitabine; Oxaliplatin

ARMS (1):
- no arms (Other): no arms were present for the study, only 2 different cohorts:MCL and LDCGB
  Interventions: Drug: Rituximab, Gemcitabine, Oxaliplatin, Dexametasone

INTERVENTIONS:
Drug: Rituximab, Gemcitabine, Oxaliplatin, Dexametasone — until progression or unacceptable toxicity develops, 8 cicles max Rituximab: 375 mg/m2, IV, day 1. Gemcitabine: 1000 mg/m2, IV, day 2. Oxaliplatin: 100 mg/m2, IV, day 2. Dexametasone: 20 mg/day, days 1-3, oral.

SUMMARY:
The purpose of this study is to determine efficacy of rituximab, gemcitabine, oxaliplatin and dexametasone (R-GemOx) chemotherapy schedule.

DETAILED DESCRIPTION:
The purpose of this study is to determine efficacy (overall response rate (ORR) and complete response) tolerance and toxicity of rituximab, gemcitabine, oxaliplatin and dexametasone (R-GemOx) chemotherapy schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. DLBCL and MCL diagnosed patients in primary resistance or relapsed not eligible for intensification chemotherapy followed by Autologous stem cell transplantation (ASCT) for age, comorbidity or previous ASCT.
3. Any IPI or ECOG, capable of understanding the nature of the trial.
4. Writtern Informed Consent.

Exclusion Criteria:

1. Nursing pregnant or lactation period women, or fertile age adults not using effective contraceptive method.
2. CNS lymphoma patients.
3. Patients with severa renal (creatinine> 2,5 UNL) or hepatic (Bilirrubin or ALT/AST> 2,5 UNL) impairement not provided by the same disease
4. HIV positive patients.
5. Serious psychiatric diseases patients that could interfere with their skill to understand the study (including alcoholism or drug addiction).
6. Murine proteins or any other component of the medicines of the study hypersensitivity patients.
7. Patients who have received more than 2 therapeutic previous lines. (for previous ASCT patients, induction and conditioning for the TAPH treatment is considered a single line therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to evaluate Overall response rate (ORR) | 3 years and 2 months
  The primary endpoint is to evaluate the number of patients with complete remission, unconfirmed complete remission and partial response according to International Workshop to Standardize Response Criteria for NHL, of R-GEMOX combination administered every 14 days

SECONDARY OUTCOMES:
Safety of Gemcitabine in combination with Rituximab, Oxaliplatin and Dexametasone (R-GemOx) in DLBCL and Mantle cell lymphoma. (GELTAMO-RGemOx) | 3 years and 2 months
  To asses the number of Participants with Adverse Events (serious and non serious) and classification of those adverse events.
  Evaluate if the balance efficacy / toxicity allows the possibility of further interventions to prolong progression-free survival and overall survival
To identify clinical response predictive factors | 3 years 2 months
  To asses if different age, sex, IPI, ECOG, stage of cancer, dissease location and time to relapse have some influence in response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés López Hernández, MD, Principal Investigator — Hospital Vall d´Hebrón; Mª Dolores Caballero Barrigón, MD, Principal Investigator — Hospital Clínico de Salamanca; Jorge Gayoso Cruz, MD, Principal Investigator — Hospital Universitario Gregorio Marañón; Juan Alfonso Soler Campos, MD, Principal Investigator — Corporació Sanitari Parc Taulí; Carlos Montalbán Sanz, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Juan Manuel Sancho Cía, MD, Principal Investigator — Germans Trias i Pujol Hospital; Isidro Jarque, MD, Principal Investigator — Hospital La Fe de Valencia; Secundino Ferrer, MD, Principal Investigator — Hospital Dr. Peset; Carlos Grande, MD, Principal Investigator — Hospital 12 de Octubre; Pilar Martínez Barranco, MD, Principal Investigator — Fundación Hospital de Alcorcón; Miguel Ángel Canales Albendea, MD, Principal Investigator — Hospital La Paz; Jose Antonio García Marco, MD, Principal Investigator — Hospital Puerta de Hierro de Majadahonda; Roberto Hernández Martín, MD, Principal Investigator — Hospital Virgen de la Concha; José Manuel Calvo Villas, MD, Principal Investigator — Hospital Dr. Jose Molina Orosa; Miguel Hernández, García, Principal Investigator — Hospital Universitario de Canarias; Elena Pérez Ceballos, MD, Principal Investigator — Hospital Morales Meseguer; José M. Moraleda Jiménez, MD, Principal Investigator — Hospital Virgen de la Arrixaca; Eulogio Conde García, MD, Principal Investigator — Hospital Marqués de Valdecilla; Carlos Panizo Santos, MD, Principal Investigator — Clínica Universitaria Navarra; Mª Rosario Varela, MD, Principal Investigator — Complejo Hospitalario A Coruña; Jose Luis Bello López, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago; Maria José Ramírez Sánchez, MD, Principal Investigator — Hospital del SAS Jerez; Luis Palomera, MD, Principal Investigator — Hospital Clínico Lozano Blesa; Pilar Giraldo, MD, Principal Investigator — Hospital Miguel Servet; Antonio Gutiérrez, MD, Principal Investigator — Hospital Son Espasses; Joan Bargay Leonart, MD, Principal Investigator — Hospital Son Llàtzer; Eva González Barca, MD, Principal Investigator — Hospital Duran i Reynals; Javier Briones Meijide, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (28):
- Spain (28):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Duran i Reynals, Sabadell, Barcelona
  - Hospital SAS de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Dr. Jose Molina Orosa, Arrecife, Lanzarote
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Virgen de Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario de A Coruña, A Coruña
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital 12 Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Morales Meseguer, Murcia
  - Hospital Son Espasses, Palma de Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Corporació Sanitari Parc Taulí, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Dr. Peset, Valencia
  - Hospital La Fe, Valencia
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza